CLINICAL TRIAL: NCT04826913
Title: High Throughput Screening Device Based on 3D Nano-matrices and 3D Tumors With Functional Vascularization
Acronym: TUMOVASC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8036
Record Dates: First submitted 2021-03-22; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: NSCLC
Keywords: organoids; drug testing; immunotherapy
MeSH Terms: interventions — Microphysiological Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * whole blood (2 sample of blood collected prior to surgery)
  * tumoral tissue (non small cell lung cancer)
  * lung tissue with no malignity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Organoids — Use of an innovative device to improve the management of patients with NSCLC for precision medicine.
  The different drugs used can be conventional chemotherapy (cisplatin, carboplatin, pemetrexed), targeted therapies or immunotherapy molecules. It is also planned to use radiotherapy on our drug testing device.

SUMMARY:
Almost 85% of new therapeutic molecules are abandoned before the clinical trial stage. Most of these failures currently concern cancer therapies.

In order to optimize the development of these molecules and allow the development of precision medicine, an innovative screening device that is as close as possible to in vivo is necessary.

For this reason, the platform the investigators are setting up takes into account tumor vascularization as well as the 3D microenvironment.

The platform the investigators intend to set up is based on 4 cornerstones:

* the formation of patient-derived organoids seems to be the best option to take into account the microenvironment and cellular interactions.
* the vascular network: the formation of a peri-tumoral vascular network, either by using HUVECS cells or by using endothelial cells from the patient.
* the extracellular matrix, and the set of proteins it contains, is a major element of in vivo interaction. Moreover, the presence of a matrix is a key element for the development of vascularization in vitro.
* Functional tumor microenvironment: peri-tumor vascularization is necessary but not sufficient to claim to recreate a tumor microenvironment. It must be functionalized, and this implies the use of a microfluidic system.

This ready-to-use platform will be used on tumor biopsies of the patient, to constitute a tool for personalized medicine. This could even be a future component of decision at multidisciplinary board meetings.

The main objective of our research is the constitution of organoids derived from the patient in order to select, via a screening device, the best anti-tumor therapy to administer to the patient.

A secondary objective is to collect lymphocytes from the patient's blood in order to test the effectiveness of therapies mediated by the immune system (immunotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years old
* Patient with non-small cell bronchopulmonary cancer (NSCLC), at any stage, undergoing surgery in the Thoracic Surgery Department of the New Civil Hospital, Strasbourg.
* Patient who agreed to participate in this observational study.
* Patient affiliated to a social security system

Exclusion Criteria:

* Refusal to participate in the study
* Known hepatitis, known HIV
* Subject under safeguard of justice
* Subject under guardianship or trusteeship
* Inability to give informed information about the subject (subject in an emergency situation, difficulties in understanding the subject)
* Pregnant Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with non-small cell bronchopulmonary cancer (NSCLC), at any stage, undergoing surgery in the Thoracic Surgery Department of the New Civil Hospital, Strasbourg.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Testing of anti-cancer drugs | 3 years
  Obtaining organoids from healthy tissue and tumor tissue. The tests will used these organoids

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided